CLINICAL TRIAL: NCT05297799
Title: Clinical Validation of the Ameda Pearl Breast Pump
Brief Title: Clinical Validation of the Ameda Pearl - An Electric, Hospital Grade, Multi-User Breast Pump
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ameda, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HGP2022
Record Dates: First submitted 2022-02-26; First posted 2022-03-28 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Breast Pumping
MeSH Terms: conditions — Breast Milk Expression

STUDY DESIGN:
Intervention Model Description: Lactating women
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Lactating women (Experimental): New mothers whose infants born after 28 weeks gestational age are unable to breastfeed will exclusively breast pump their breast milk with an Ameda Pearl breast pump for a minimum of the first 14 days postpartum.
  Interventions: Device: Ameda Pearl breast pump

INTERVENTIONS:
Device: Ameda Pearl breast pump — The Ameda Pearl breast pump is a powered, multi-user breast pump with stimulation and expression modes and independently user-selectable speed and suction control in each mode.

SUMMARY:
This study introduces a new Ameda electric multi-user, hospital-grade breast pump, the Ameda Pearl, to mothers who choose to exclusively breast pump until their infants are able to breastfeed.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether exclusively pumping mothers of hospitalized infants greater than or equal to 28 weeks gestational age can come to volume, defined as a minimum of 500ml/24 hours, while using the Ameda Pearl breast pump during the first 14 days postpartum.

The Ameda Pearl has a stimulation and expression mode, as well as separate speed (30-120 cycles per minute) and suction (-30 to -250 mmHg) push-button controls that are adjustable in each mode.

Study data will include daily milk volumes, suction pressures, pumping times, ending speeds and comfort by mothers of preterm infants to determine if the pump facilitates achievement of 'coming to volume' status.

ELIGIBILITY:
Inclusion Criteria:

* Delivered an infant >28 weeks gestational age
* Infant is unlikely to be developmentally ready to breastfeed until >2 weeks old
* Wish to initiate lactation and express breast milk for at least two weeks, exclusively using the study pump
* Started or plan to start pumping within six hours of delivery
* Agree to double pump with study pump to express breast milk at least 8 times per 24 hours for a minimum of 15 minutes each session during the study participation period
* Read and understand the English language
* Adults, over or equal to the age of 18 are being recruited in this study so consent can be given by the participant directly. These potential participants could be included in the study if their infants were born in the third trimester, greater than or equal to 28 weeks gestational age, and were unable to breastfeed due to prematurity, developmental stage and/or physical anomalies preventing their ability to breastfeed directly at the breast.

Exclusion Criteria:

* Have had breast reduction surgery
* Have a history of low milk production
* Have any medical or physical condition that in the opinion of the investigator would prevent them from participating in the study
* Are currently breastfeeding another child
* Fail the initial Investigator Breast Tissue Assessment (Attachment #4)
* Have begun breast pumping with another breast pump to express breast milk
* Are taking any medications or supplements that are meant to alter milk supply volume

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-07-21 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
milk volume | At day 14
  milk volume pumped during multiple sessions over a 24-hour period

CONTACTS AND LOCATIONS:
Overall Officials: Susan M Shondel, MD, Principal Investigator — Summa Health
Locations (1):
- Summa Health, Akron, Ohio, United States

IPD SHARING:
Plan to Share IPD: No